CLINICAL TRIAL: NCT00708565
Title: Effects of Iloprost on Hypoxic Pulmonary Vasoconstriction and Exercise Capacity at High Altitude
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: VA Loma Linda Health Care System (U.S. Federal Agency)
Collaborators: Actelion (Industry)
Responsible Party: James D Anholm, MD, VA Loma Linda Healthcare System
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 00769
Record Dates: First submitted 2008-06-30; First posted 2008-07-02 (Estimated); Last update posted 2008-07-02 (Estimated); Status verified 2008-06

CONDITIONS: Hypoxic Pulmonary Vasoconstriction
Keywords: To study the effects of iloprost on hypoxic pulmonary vasoconstriction at high altitude
MeSH Terms: interventions — Iloprost

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: iloprost — Baseline echo measurements, cardiac output, pulse oximetry will be taken. Subjects will then be given one dose of inhaled iloprost. Post-inhalation, the measurements will be repeated at rest and with exercise.
  Other Names: Ventavis (brand name)

SUMMARY:
The objective of this study is to determine if single dose administration of inhaled iloprost will reduce pulmonary artery pressure, reduce hypoxic pulmonary vasoconstriction and improve arterial oxygenation at rest and during exercise at high altitude.

DETAILED DESCRIPTION:
Three major pathways in addition to oxygen modulate pulmonary vascular tone: 1) nitric oxide, 2) endothelin, and 3) prostacyclin. Considerable animal data support the role of the prostacyclin pathway in modulating hypoxic pulmonary vasoconstriction. In humans, prostacyclin and its analogs are important therapeutic agents in the treatment of pulmonary arterial hypertension (PAH). Despite the animal data and human data in PAH there is very little information about the use of iloprost to relieve hypoxic pulmonary vasoconstriction in healthy humans. Inhaled iloprost is an ideal agent to study the prostacyclin pathway due to its short duration of action (30-90 min) and elimination half-life of only 20-30 min. Individuals already participating in the Nepal Medex 2008 trip will be invited to participate in this research. Participants will be healthy active females or males, between 18-80 years of age, without known pregnancy or liver disease, who have a readily measurable tricuspid regurgitant velocity by Doppler echocardiography. If possible, we will attempt to identify a cohort of HAPE susceptible patients. Participants will undergo evaluation both at sea level (baseline) and at high altitude. Baseline (low altitude) testing will be performed in Bangor, North Wales, UK, and will include evaluation of pulmonary artery systolic pressures, cardiac output, and oxygen saturation at rest and during submaximal exercise before and after inhalation of iloprost. This strategy will then be repeated at an altitude of approximately 5000 meters in the Dhaulagiri region of Nepal.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18 - 80 years
2. Healthy physically active males or females
3. Have readily measurable tricuspid regurgitation (TR) peak systolic velocity by continuous wave Doppler ultrasound

Exclusion Criteria:

1. Unable to measure TR velocity
2. Known liver disease
3. Pregnancy
4. Nitrates, cyclosporin, glyburide or other medications that in the opinion of the investigators could place subjects at increased risk of complications
5. Any other medical condition that in the opinion of the investigators would place the subject at high risk

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2008-07; Primary Completion 2008-10 (Estimated); Study Completion 2008-10 (Estimated)

PRIMARY OUTCOMES:
Exercise capacity, pulmonary artery systolic pressure, cardiac output, oxygen saturation | 6 months

SECONDARY OUTCOMES:
Heart rate, tissue Doppler echocardiographic measurements | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: James D Anholm, MD, Principal Investigator — Jerry L. Pettis VA Mecial Center
Locations (1):
- Jerry L. Pettis VA Medical Center, Loma Linda, California, United States